CLINICAL TRIAL: NCT05809609
Title: Does Modulation of Glutamate Transmission in the Brain Using a Sub-anaesthetic Dose of Ketamine Affect Autobiographical Memory, Emotional Processing and Decision-making in Treatment-resistant Depression?
Brief Title: Glutamate Emotion Memory Study
Acronym: GEMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GEMS
Record Dates: First submitted 2022-04-26; First posted 2023-04-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Treatment Resistant Depression; Depression; Major Depressive Disorder
Keywords: Ketamine; Memory; Mental Health; Learning
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Depressive Disorder, Major; Psychological Well-Being | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive ketamine or placebo. Ketamine is not being administered for treatment purposes, the purpose is to understand the mechanisms underpinning its effects.
Who Masked: Participant, Investigator
Masking Description: All members of the study team will be blinded to the condition a participant is allocated to with the exception of the team member responsible for administering the drug/placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants in this arm will receive a single intravenous injection, antidepressant dose of Ketamine hydrochloride (0.5mg/kg)
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): Participants in this arm will receive a single intravenous injection of an inactive placebo (0.9% sodium chloride)
  Interventions: Other: No intervention (placebo)

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine is a high trapping NMDA receptor antagonist which has rapid and reliable antidepressant effects in patients with major depressive disorder (MDD) who fail to respond to at least two antidepressant trials of adequate dose and duration.
  Arms: Ketamine
Other: No intervention (placebo) — Placebo injection (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
Clinical depression often includes a pessimistic view of things which have happened in the past and an impairment in the ability to experience pleasure or looking forward to things. A licensed drug called ketamine affects the levels of glutamate, a chemical messenger in the brain, and has been used as a treatment particularly for depression which hasn't got better with other types of medication. Glutamate plays a role in learning and memory so the investigators are interested in understanding how ketamine can affect how people with depression remember past negative and positive memories and how they experience reward.

The investigators are conducting a study in depressed participants who did not improve with the standard antidepressant treatment to expand our understanding on how ketamine can influence memory, the way people understand emotions and learn from rewards and punishments. Study participants will undergo medical and psychiatric health screening, drug administration (ketamine or saline), questionnaires and computer tasks before and after the administration of the study drug, and an MRI scan after administration of the drug. MRI is a type of brain scan that allows us to see how the brain responds during for example memories of things which have happened in the past. This project will help us understand how NMDA antagonists may work in depression.

DETAILED DESCRIPTION:
Questions regarding the exact molecular mechanisms of ketamine and its effects on the brain circuitry and networks for the treatment of clinical depression remain largely unanswered. Thus, in the present study the investigators aim to elucidate the effect of ketamine on 1) reconsolidation of autobiographical memories, 2) connectivity of brain circuits involved in autobiographical memories, 3) measures of emotional processing, reward processing and emotional memory in patients suffering from treatment resistant depression. The ultimate goal of this project is to elucidate the antidepressant mechanisms of action of ketamine to facilitate the development of rapid acting antidepressants targeting the glutamatergic system.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Sufficiently fluent English to understand and complete the tasks
* Registered with a GP and consents to GP being informed of participation in the study

Participants need to meet a number of concurrent clinical criteria:

* Current criteria for Major Depressive Disorder, in a current major depressive episode as determined by the SCID-5.
* Inadequate response to at least one and no more than three antidepressant treatments.
* Currently taking a licensed antidepressant at a therapeutic dose for at least four weeks.
* Pre-menopausal women and male participants engaging in sex with a risk of pregnancy must agree to use a highly effective method of contraception from Screening Visit until 30 days after receiving the study medication treatment.

Acceptable methods of contraception include:

* Condoms
* Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation oral, injectable or implantable
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomy (or vasectomised partner)
* Sexual abstinence. [Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), and spermicides only are not acceptable methods of contraception.]
* Male participants must not donate sperm until 30 days after receiving the study medication.
* Participants taking non-prescription/prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety
* Willingness to refrain from driving, cycling, or operating heavy machinery, until the following morning or a restful sleep has occurred, whichever is later.
* Willingness to refrain from drinking alcohol for 3 days before the infusion visit and one day before any of the other visits throughout the study.

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:
* History of /or current DSM-5 bipolar disorder, schizophrenia or emotionally unstable personality disorder [co-morbid anxiety disorders (including agoraphobia, generalized anxiety disorder, social anxiety disorder and panic disorder) and Posttraumatic Stress Disorder (PTSD) are allowed]
* Participants who fulfil current criteria for other comorbid disorders may still be entered into the study, if, in the opinion of the Investigator, the psychiatric diagnosis will not compromise safety or affect data quality
* Diagnosis of a major cognitive disorder or evidence of cognitive impairment
* Clinically significant risk of suicide
* Participants undergoing or who have undergone electroconvulsive therapy for the treatment of the current episode of depression
* Substance or alcohol use disorder over the past 6 months
* Regular alcohol consumption of more than 21 units a week or excessive alcohol consumption up to three days before any of the in-person study visits or inability to abstain from alcohol for more than 3 days
* Moderate cigarette use (> 10 cigarettes per day)
* History of, or current general medical conditions that in the opinion of the Investigator may interfere with the safety of the participant or the scientific integrity of the study
* Current pregnancy (as determined by urine pregnancy test), breastfeeding, planning a pregnancy, or unwillingness to practice birth control during the course of the study
* Clinically significant abnormalities of laboratory tests, physical examination, or ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Current or past history of heart rhythm disorders
* Clinically significant untreated hypertension
* Any contraindication to MRI including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more
* Previous participation in a study using the same, or similar, emotional processing tasks in the last three months
* Previous lifetime use of ketamine or phencyclidine
* Participant with planned medical treatment within the study period that might interfere with the study procedures
* Participant who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in magnitude of negative and positive valence adjectives in the autobiographical memory task using a self-reported questionnaire. | -1 and 1 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - negative emotional bias associated with autobiographical memories in TRD patients.
  Each negative (guilty/ashamed, depressed/sad, angry/frustrated, upset, anxious/worried, worthless) and positive (grateful, energetic/motivated, hopeful, confident, loved, happy) valence adjectives. will be rated on a scale from 0 to 100. Change in magnitude will be assessed calculating the difference in ratings of negative and positive adjectives using a self-reported questionnaire from baseline to after treatment
Brain activation as measured by functional magnetic resonance in a network of areas related to autobiographical memories, including the medial prefrontal cortex and associated networks during the autobiographical memory task. | 1 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - on brain circuit associated with autobiographical memories

SECONDARY OUTCOMES:
Accuracy on a computer-based task of facial expression recognition (FERT) | -1 day, and up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as emotional recognition.
Reaction time on a computer-based task of facial expression recognition (FERT) | -1 day, and up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as emotional recognition.
Accuracy to classify positive and negative descriptor words using the Emotional Categorisation Task (ECAT) | Up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as classification of positive and negative descriptor words
Reaction time to classify positive and negative descriptor words using the Emotional Categorisation Task (ECAT) | Up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as classification of positive and negative descriptor words
Number of positive and negative words correctly recalled (hits) and number of words incorrectly recalled (false alarms) using the Emotional Recall Task (EREC) | Up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as recall of positive and negative descriptor words
Accuracy to correctly (hits) and incorrectly (false alarms) recognise positive and negative words using the Emotional Recognition Memory Task (EMEM) | Up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as recognition of positive and negative descriptor words
Reaction time to correctly (hits) and incorrectly (false alarms) recognise positive and negative words using the Emotional Recognition Memory Task (EMEM) | Up to 2 hours after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - emotional processing such as recognition of positive and negative descriptor words
Change in response choice during gain and loss using the Probabilistic Instrumental Learning Tasks (PILT) | 1 day after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - reward processing
Brain activation as measured by functional magnetic resonance imaging during the Probabilistic Instrumental Learning Tasks (PILT) in reward-related brain areas, including the ventral striatum and associated networks | 1 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - on brain circuit associated with reward processing
Explore performance on information processing and monetary win/loss reinforcement learning (RL) decision-making tasks. | 1 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - choice behaviour on win and loss trials
Explore performance on information processing and monetary win/loss reinforcement learning (RL) decision-making tasks using pupillometry | 1 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - pupil dilation in context of RL decision making task
Change in choice behaviour (effort and/or reward sensitivity) on accepted offers between session one and two using the Apples Gathering Task (AGT). | Up to 2 hours after ketamine/placebo treatment and 7 days after ketamine/placebo treatment
  To investigate the effects of ketamine on:
  - motivation processing

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, United Kingdom